CLINICAL TRIAL: NCT06166654
Title: Optimal Diuretic Therapies for Acute Heart Failure With Volume Overload - A Randomized Clinical Trial
Brief Title: Optimal Diuretic Therapies for Acute Heart Failure With Volume Overload
Acronym: DRAIN-AHF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johannes Grand (Other)
Responsible Party: Sponsor-Investigator, Johannes Grand, Principal Investigator, Copenhagen University Hospital, Hvidovre
Organization: Copenhagen University Hospital, Hvidovre (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRAIN_AHF
Record Dates: First submitted 2023-12-03; First posted 2023-12-12 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Acute Heart Failure
Keywords: acute heart failure; decongestion; diuretic
MeSH Terms: interventions — Acetazolamide; Metolazone

STUDY DESIGN:
Intervention Model Description: 3-arm parallel group RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will employ a triple-blind design (Participants and relatives, investigators and clinicians, and data analysts and outcome adjudicators)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acetazolamide (Active Comparator): 1. 500 mg IV bolus of acetazolamide at randomization (day 0) and repeated the next 3 mornings (day 1, day 2 and day 3). This arm will also receive a placebo- Metolazone tablet together with each acetazolamide-injection.
  Interventions: Drug: Acetazolamide
- Metolazone (Active Comparator): 2.5 mg oral Metolazone at randomization (day 0) and repeated the next 3 mornings (day 1, day 2 and day 3). This arm will also receive a placebo- acetazolamide injection together with each metolazone-tablet.
  Interventions: Drug: Metolazone 2.5 MG
- Placebo (Placebo Comparator): Usual care with loop-diuretics as the sole diuretic (SGLT2-inhibitors allowed) including guideline-recommended increase in loop-diuretic dose and fluid and salt-restriction. This arm will also receive both a placebo-acetazolamide injection together with a placebo-metolazone-tablet at randomization and repeated the next 3 mornings (day 1, day 2 and day 3).
  Interventions: Other: Double-placebo

INTERVENTIONS:
Drug: Acetazolamide — 1. 500 mg IV bolus of acetazolamide at randomization (day 0) and repeated the next 3 mornings (day 1, day 2 and day 3). This arm will also receive a placebo- Metolazone tablet together with each acetazolamide-injection.
  Other Names: Standard of care including loop-diuretics
  Arms: Acetazolamide
Drug: Metolazone 2.5 MG — 2. 2.5 mg oral Metolazone at randomization (day 0) and repeated the next 3 mornings (day 1, day 2 and day 3). This arm will also receive a placebo- acetazolamide injection together with each metolazone-tablet.
  Other Names: Standard of care including loop-diuretics
  Arms: Metolazone
Other: Double-placebo — This arm will also receive both a placebo-acetazolamide injection together with a placebo-metolazone-tablet at randomization and repeated the next 3 mornings (day 1, day 2 and day 3).
  Arms: Placebo

SUMMARY:
Aim to identify the best strategy for treating acute heart failure (AHF) with volume overload, particularly focusing on patients resistant to standard loop-diuretics. The trial is a double-blinded, randomized, controlled, multicenter study. Its primary objective is to compare the efficacy of loop-diuretics combined with either Metolazone or Acetazolamide, against loop-diuretics alone. The trial will also determine the optimal type of loop-diuretic to use.

Eligible participants include adults over 18 years hospitalized with AHF and volume overload, showing signs of congestion and at risk of diuretic resistance. Exclusions apply to those with acute coronary syndrome, low systolic blood pressure, prior renal therapy, or previous treatment with Acetazolamide or Metolazone.

The primary outcome is the number of days alive and out-of-hospital by day 30. Secondary outcomes include a composite clinical benefit at 30 days, Kansas City Cardiomyopathy Questionnaire (KCCQ) scores, and successful decongestion 72 hours post-inclusion.

The trial aims to enroll about 1,041,939 patients across three treatment arms over three years. The minimal important difference is set as a reduction in out-of-hospital days by at least two days, with an anticipated low dropout rate. The study's power is calculated to be 80% with an adjusted alpha level for comparing the three diuretic groups.

DETAILED DESCRIPTION:
Trial synopsis Title: OPTIMAL DIURETIC THERAPIES FOR ACUTE HEART FAILURE WITH VOLUME OVERLOAD - A RANDOMIZED CLINICAL TRIAL

Background:

Intravenous loop-diuretics have been the key component in treating acute heart failure (AHF) since the nineteen sixties and has a Class 1 recommendation in the 2021 ESC guidelines for heart failure. Hospitalization for AHF with volume overload is the most frequent cause of hospital admission among elderly patients and is associated with poor outcome. There is a high need for additional decongestant therapies beyond the recommended use of intravenous loop diuretics.

Primary objective:

To determine the superior strategy of loop-diuretics + Metolazone, loop-diuretics + Acetazolamide, or loop-diuretics without additional diuretics during in-hospital treatment for acute decompensated heart failure with volume overload and diuretic resistance. Furthermore, to determine optimal type of loop-diuretic.

Hypothesis:

One of the three diuretic strategies are superior to the others for decongesting acute heart failure with volume overload.

Design: Investigator-initiated, double-blinded, randomized, controlled, multicenter, interventional clinical trial of acute decompensated heart failure patients at risk for diuretic resistanseresistance.

Intervention:

* Acetazolamide as add-on to loop-diuretics
* Metolazone as add-on to loop diuretics
* Usual care including guideline-recommended increase in loop-diuretic dose and fluid and salt-restriction.

Inclusion criteria:

1. Age ≥ 18 years
2. Acute hospital admission with a clinical diagnosis of acute heart failure with volume overload.
3. At risk of diuretic resistance
4. Clinical signs of congestion

Exclusion criteria:

1. Acute coronary syndrome
2. Systolic blood pressure <85 mmHg
3. Use of renal replacement therapy or ultrafiltration in-hospital before study inclusion
4. Treatment with acetazolamide or metolazone during hospitalization prior to randomization

Primary outcome: Days alive out-of-hospital to day 30.

Secondary outcomes:

1. Clinical benefit at 30 days, consisting of a composite of 1. all-cause death, 2. Readmisison after discharge from initial hospitalization, 3. new receipt of renal-replacement therapy, or persistent renal dysfunction (defined as a final inpatient creatinine value ≥200% of the baseline value), assessed using a Hierarchical win-ratio' approach.
2. Kansas City Cardiomyopathy Questionnaire (KCCQ) at 30 days
3. Successful decongestion 72 hours after inclusion (measured as the decongestion score ad modum Advor)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Acute hospital admission with a clinical diagnosis of acute heart failure with volume overload.
3. Display risk of diuretic resistance, characterized by:

   1. Daily loop-diuretics administration for a minimum of 7 days before admission, or
   2. Insufficient decongestion observed in the preceding 24 hours (weight reduction <500g or negative fluid balance <1L) despite being treated with high-dose IV loop diuretic (equivalent to ≥120 mg IV furosemide within 24 hours).
4. Clinical signs of congestion, indicated by one or more of the following: pitting peripheral edema, ascites, elevated jugular venous pressure, or radiological/ultrasonic evidence of pulmonary congestion.

Exclusion Criteria:

1. Acute coronary syndrome
2. Systolic blood pressure <85 mmHg
3. Use of renal replacement therapy or ultrafiltration in-hospital before study inclusion
4. Treatment with acetazolamide or metolazone during the index hospitalization prior to randomization
5. Known allergy to any of the used drugs
6. Severe hypokalemia (<2.5 mmol/l) or severe hyponatremia (<125 mmol/l)
7. Severe hepatic impairment or liver cirrhosis
8. Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 939 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Days alive out-of-hospital to day 30 | 30 days
  Days alive out-of-hospital to day 30

SECONDARY OUTCOMES:
Win ratio of 1. all-cause death, 2. Readmisison, 3. renal-replacement therapy, or persistent renal dysfunction (defined as a final inpatient creatinine value ≥200% of the baseline value), assessed using a Hierarchical win-ratio' approach. | 30 days
  Number of Clinical benefit at 30 days, consisting of a composite of 1. all-cause death, 2. Readmisison after discharge from initial hospitalization, 3. new receipt of renal-replacement therapy, or persistent renal dysfunction (defined as a final inpatient creatinine value ≥200% of the baseline value), assessed using a Hierarchical win-ratio' approach.
Kansas City Cardiomyopathy Questionnaire | 30 days
  Kansas City Cardiomyopathy Questionnaire (KCCQ). Minimum and Maximum Values: The KCCQ is scored on a scale from 0 to 100.
  Interpretation of Scores:
  Higher Scores: Indicate better heart failure-related quality of life, fewer symptoms, and fewer physical and social limitations.
  Lower Scores: Suggest more severe heart failure symptoms, greater physical limitations, and a poorer quality of life.
Decongestion score 72 hours after inclusion | 72 hours
  scale from 0 to 10 on the basis of the sum of scores for the degree of edema (0 to 4), pleural effusion (0 to 3), and ascites (0 to 3), with higher scores indicating a worse condition on all scales

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Grand, MD, Phd, MPH, Principal Investigator — Amager-Hvidovre Hospital
Locations (3):
- Denmark (3):
  - Amager-Hvidovre Hospital, Hvidovre, Capital Region of Denmark
  - Bispebjerg Hospital, Copenhagen
  - Herlev-Gentofte hospital, Copenhagen

IPD SHARING:
Plan to Share IPD: No